CLINICAL TRIAL: NCT06549205
Title: Effects of Trigeminal Neurostimulation on Heart Rate Variability: Comparing Cutaneous (Tragus) and Tongue (Antero-Dorsal Mucosa) Stimulation.
Brief Title: Effects of Trigeminal Neurostimulation on Heart Rate Variability: Comparing Tragus and Tongue Stimulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Sara Di Nicolantonio, PhD candidate, University of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16137/2016
Record Dates: First submitted 2024-08-01; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Arousal, Confusional
Keywords: Trigeminal electrical stimulation; ULFTENS; Heart rate variability; tragus; tongue
MeSH Terms: conditions — Sleep Arousal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUD group (Experimental): an intraoral device will be administered in the TUD group in order to provide the stimulation of the dorsal surface of the tongue with dental TENS. The trial will last approximately 24 minutes, after the first 6 minutes, TENS activation will take place and how HRV values change will be evaluated. The Heart rate Variability parameters will be analysed with photopletismographic wave after 6 minutes of tongue stimulation
  Interventions: Device: device that stimulates the dorsal surface of the tongue
- Tragus group (Active Comparator): patients in this group will be administered traditional trigeminal stimulation with dental TENS at tragus level. Tens will be turned on for 6 minutes in which the HRV parameters will be analyzed with the photoplethysmograph and compared with the data obtained in the TUD group.
  Interventions: Device: device that stimulates the tragus

INTERVENTIONS:
Device: device that stimulates the dorsal surface of the tongue — the device will be placed on the dorsal surface of the tongue. this instrument has two electrodes in turn connected to the TENS, so ultra low frequency stimulation (<0.66 Hz) will be administered
  Arms: TUD group
Device: device that stimulates the tragus — two electrodes will be placed at tragus level for the administration of dental ULFTENS
  Arms: Tragus group

SUMMARY:
this study wants to analyse the effect of trigeminal stimulation on Heart rate Variability. There are going to be two groups, in the test group it will be administered stimulation of the tongue with TENS, while in the control goup TENS will be administered at tragus level.

DETAILED DESCRIPTION:
This study analyses the effect of trigeminal stimulation with TENS on Heart rate variability (HRV). A new intraoral device will be administered on the dorsal surface of the tongue for TENS stimulation in the test group. The RMSSD, LF, HF and LF/HF will be monitered by photoplethysmographic wave. the results obtained with tongue stimulation will be compared with the results obtained in the control group, where it will be administered TENS stimulation at the tragus level. This work sought to assess whether there is a difference in HRV in relation to the site of application of dental ULFTENS (tragus vs tongue).

If effective in reducing the activity of arousal circuits, this tongue-level stimulation technique could have new clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Women
* Age 18-30 years

Exclusion Criteria:

* presence of acute and/or chronic cardio-circulatory and respiratory disorders
* metabolic and autonomic system disorders
* intake of excitatory or inhibiting substances of the peripheral and central nervous system
* presence of generalised anxiety and/or panic attacks or mood disorders.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Changes on Low Frequency parameter (LF) | 12 minutes
  Whether or not HRV parameter (LF) improve following tongue and tragus stimulation will be assessed by photopletismographic wave
Changes on Root mean square standard deviation (RMSSD) parameter | 12 minutes
  Whether or not HRV parameter (RMSSD) improve following tongue and tragus stimulation will be assessed by photopletismographic wave

CONTACTS AND LOCATIONS:
Locations (1):
- Sara Di Nicolantonio, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monaco A, Cattaneo R, Di Nicolantonio S, Strada M, Pietropaoli D, Ortu E. Effects of trigeminal neurostimulation on heart rate variability: comparing cutaneous (Tragus) and tongue (Antero-Dorsal mucosa) stimulation. BMC Oral Health. 2024 Oct 20;24(1):1257. doi: 10.1186/s12903-024-04914-2. PMID 39428464

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT06549205/Prot_SAP_ICF_000.pdf